CLINICAL TRIAL: NCT04926519
Title: Periodontitis in Young Individuals, Follow up of Treatment and Disease Progression Over 10 Years
Status: Completed | Type: Observational
Sponsor: Folktandvården Stockholms län AB (Other Government)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Carolina Modin, DDS, Senior Consultant in Periodontology, Folktandvården Stockholms län AB
Other Study IDs: 556574-3597
Record Dates: First submitted 2020-10-02; First posted 2021-06-15 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Periodontitis
Keywords: severe periodontitis; long-term disease progression
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Bacterial samples from deep periodontal pockets and samples of gingival crevicular fluid from deep periodontal pockets
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Aggressive periodontitis: Patients that got the diagnosis aggressive periodontitis at baseline. Since 2018 we have the classification system with stage and grade why patients get this classification at the clinical examination.
  Interventions: Other: Type of periodontal treatment
- Chronic periodontitis: Patients that got the diagnosis chronic periodontitis at baseline. Since 2018 we have the classification system with stage and grade why patients get this classification at the clinical examination.
  Interventions: Other: Type of periodontal treatment

INTERVENTIONS:
Other: Type of periodontal treatment — Identify factors that contribute to disease recurrence due to periodontal classification and periodontal treatment. One group have got the diagnosis aggressive periodontitis at baseline and the other group chronic periodontitis. Since 2018 we have the classification system with stage and grade.

SUMMARY:
The general aim of this project is to get a better understanding how periodontitis develop in young individuals over time and identify factors that contribute to disease recurrence. The investigators also want to see if Stage and Grade of the periodontal disease has a significant impact on disease progression. In addition, another purpose is to identify factors explaining why certain young patients with periodontitis interrupt the periodontal treatment.

The specific aims of the project are:

* To study the periodontal status and the degree of disease progression over 10 years for young individuals with periodontitis at age < 36 yrs at baseline (study 1)
* To identify factors with a significant influence on periodontitis progression for young individuals with periodontitis at baseline (study 2)
* To identify explanatory factors to discontinuation of periodontal treatment (study 3)
* To identify bio marker and microbiological profiles in young individuals in relation to stage and grade of periodontitis (study 4)

Significance:

A high patient compliance rate and effective supportive treatment to prevent periodontitis progression are crucial conditions for the long-term prognosis. The identification of factors influencing the compliance rate can improve the frequency of individuals following a supportive care program. In addition, long-time follow-up studies of individuals with the diagnosis severe periodontitis at young age are lacking as well as deeper knowledge concerning risk predictors for further disease progression.

The identification of biomarkers or microorganisms that can differentiate between different stage and grade of periodontitis could make it possible to identify individuals with a high risk for disease progression at an early stage.

DETAILED DESCRIPTION:
Data collection:

All patients at age <36 years who were examined by a periodontist at 2 specialist clinics in Periodontology (Folktandvården Stockholm) during the years 2003-2009 with the diagnoses aggressive or chronic periodontitis are included in the project. The material consists of 471 patients. All participants are invited by mail to a clinical and radiographic examination. The clinical examination includes periodontal status and microbiological sampling and samples of crevicular fluid from deepened periodontal pockets >6. At time of examination the participants also fill in an questionnaire regarding oral hygiene habits, socio-economic factors and self-percieved oral health. Baseline information is collected from dental records.

Studies 1 and 2:

Title study 1: Periodontal status and disease progression after 10 years in young individuals with periodontitis. A follow-up study.

Title study 2: Risk predictors for periodontitis progression in young individuals with periodontitis.

Study variables:

The following variables were registered from dental records:

Diagnoses: Aggressive or chronic periodontitis, local or general periodontitis, age at baseline, sex, smoking habits at baseline, number of remaining teeth, general degree of marginal bone, presence of angular bony defects , bleeding index, periodontal pocket depths at four sites/tooth, presence of furcation involvements, mobility (degree 0-3), periodontal treatment after baseline investigation (non-surgical treatment, surgical treatment, antibiotic treatment, supportive care, treatment interrupted)

The following variables will be registered at the clinical investigation:

Number of years since baseline, number of remaining teeth, general degree of marginal bone loss, presence of angular bony defects, bleeding index, periodontal pocket depths at four sites/tooth, presence of furcation involvements, mobility (degree 0-3), microbiological test if minimum of one site bleeding on probing with periodontal pocket depth >6mm, Samples of crevicular fluid from deepened periodontal pockets >6, saliva specimens, stimulated saliva collected for two minutes

Radiografic examination: panorama x-rays and six IO x-rays

The diagnosis at baseline (chronic or aggressive periodontitis) will be transformed to the new periodontal classification system.

The following variables will be registered from a questionnaire at the clinical investigation:

Smoking habits, general health, socio-economic variables, frequency of dental visits during the follow-up period, frequency of supportive care during the follow-up period, oral hygiene habits, subjective symptoms from the mouth

Study 3:

Title: A retrospective follow-up over 10 years of dental care for young individuals with periodontitis

Study variables:

The following variables were registered from the dental records at baseline and the following treatment periods:

Year of baseline investigation, age, sex, smoking habits, general health, number of teeth at baseline, periodontal pocket depths at baseline, bleeding on probing score at baseline, tooth mobility at baseline, presence of furcation involvement at baseline, presence of angular bony defects at baseline, periodontal diagnosis, number of dental visits, treatment interrupted, number of teeth at re-evaluation, periodontal pocket depths at re-evaluation, bleeding on probing score at re-evaluation, year of the last re-evaluation.

The diagnosis at baseline (chronic or aggressive periodontitis) will be transformed to the new classification system.

The following variables will be registered from Tandhälsoregistret (register of dental health) at the National Board of Health and Welfare:

Age at dental visits, years of dental visits, country of birth, number of teeth, citizenship, date of migration, public/private dental care, marital status, kind of dental treatment, dental diagnosis, tooth number, tooth position.

Study 4:

Title: Bio marker and microbiological profiles in young individuals in relation to stage and grade of periodontitis.

Data collection: Saliva specimens are obtained by collecting unstimulated saliva for two minutes and stored at -70 degrees C until analyses. The levels of cytokines and bone resorption markers in the saliva samples will be analyzed using the Luminex technology on a Bioplex Suspension Array System (Bio-Rad Laboratories), Milliplex MAP bone metabolism kits (Millipore) or Fluorokine MAP Multiplex MMP (R&D Systems). Bacterial samples will be collected from the periodontal pockets with sterile paper points. The microbiological analyses will be performed using DNA extraction with 16S rRNA Sequencing.

Study variables:

The following cytokines will be analyzed: G-CSF, GM-CSF, IFN-gamma, IL1-β, IL-4, IL-6, IL-7, IL-8, IL-10, IL-12p70, IL-13, IL-15, IL-18, M-CSF, MIP-1α, MIP-1β, RANTES, eotaxin TNF-alfa, MCP-1, The following bone resorption markers will be analyzed: RANKL, OPG, Osteopontin, Osteocalcin, MMP-8 and MMP-9, Salivary flow, Distribution of microbiota

ELIGIBILITY:
Inclusion Criteria:

• All patients with diagnoses aggressive or chronic periodontitis

Exclusion Criteria:

* Not living in Stockholm County
* Mental illness.

Max Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All patients at age < 36 years who were examined by a periodontist at two specialist clinics in Stockholm during the years 2003-2009 (baseline) and got the diagnoses aggressive or chronic periodontitis were included in the project.
  Study group: Patients with diagnosis aggressive periodontitis at baseline Control group: Patients with diagnosis chronic periodontitis at baseline
Sampling Method: Non-Probability Sample
Enrollment: 471 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-08-15 (Actual)

PRIMARY OUTCOMES:
Periodontal disease progression in young individuals with periodontitis 10-13 years after baseline | October 2018 to May 2021
  Periodontal progression will be assessed by Periodontitis grade according to The 2017 World Workshop on the Classification of Periodontal and Peri-Implant Diseases and Conditions:
  This is a categorical variable consisting of ordinal data at three levels (A, B, C). A is the lowest progression rate and C is the highest rate.
  The assessment is performed by comparing the degree of periodontal bone loss between baseline and follow-up.

SECONDARY OUTCOMES:
Factors influencing tooth loss over 9 - 11 years in young individuals with periodontitis | 2020 to 2022
  The primary outcome variable was the number of teeth lost due to periodontitis during the follow-up period (2009-2019).
  Variables were collected from digital dental records combined with two national health registers; Swedish Dental Health register and Statistics Sweden Baseline clinical periodontal variables and information about interruption of APT at the specialist clinic (secondary outcome variable) were collected from dental records at periodontal clinics between 2003-2010.
To identify bio marker and microbiological profiles in young individuals in relation to stage and grade of periodontitis | 2020-2023
  Cytokine- and bone resorption markers:
  This is a continuous variable and the levels in the crevicular fluid are expressed as pg/ml.
  Microbiological analyses:
  We will analyse number of bacteria. Comparing healthy sites with diseased ones. This method will give us information if any of the analysed bacteria are overrepresented

CONTACTS AND LOCATIONS:
Overall Officials: Leif Jansson, DDSPhDAssPro, Principal Investigator — Folktandvården Stockholm
Locations (1):
- Folktandvården Eastmaninstitutet, Stockholm, Sweden